CLINICAL TRIAL: NCT02824289
Title: Sun Safe Workplaces: A Campaign on Sun Protection Policies for Outdoor Workers
Acronym: SSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: University of Colorado, Denver (Other); Kaiser Foundation Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA134705 (NIH)
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Skin Cancer
Keywords: skin cancer; prevention; worksite; policy
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sun Safe Workplaces Program (Experimental): Program promoting the adoption of occupational sun protection policies by the local government organization comprised of personal visits with senior managers and in-person training of outdoor workers by research staff over two years.
  Interventions: Behavioral: Sun Safe Workplaces Program
- Attention Control (Active Comparator): Program promoting occupational sun protection practices by employees in local government organizations through two mailings containing educational materials and presentations at state professional meetings by project staff.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Sun Safe Workplaces Program — The intervention began by sending a Program Announcement Packet and requesting the first face-to-face meeting. At the first meeting, intervention staff covered: 1) Introduction to SSW; 2) Sun Safety Practices in the Workplace; 3) Sun Safety Policy for Outdoor Workers; 4) Sun Safety Policy Adoption; 5) Sun Safety Policy Reinforcement and Maintenance. They presented the SSW Website and a Sun Safety Tool Box. Following the first meeting, the manager scheduled Sun Safety Training by intervention staff with various employee groups. Workplace Sun Safety Materials were sent in four sets (twice a year over two years) for distribution to employees. Research staff made monthly Follow-up Contacts with managers.
  Arms: Sun Safe Workplaces Program
Behavioral: Attention Control — Research staff sent printed materials on occupational sun safety to local government organizations twice. These included posters with personal protection messages and skin cancer rates, risk assessment brochures, worksite guides, total skin self-examination CD-Rom, the American Academy of Dermatology SPOT bookmark, and a sun safety tip card from the Occupational Safety and Health Administration (OSHA). Staff made presentations on general sun safety topics (not policy) at state professional conferences.
  Arms: Attention Control

SUMMARY:
A sample of local government organizations are recruited to a group-randomized pretest-posttest controlled trial evaluating the effect of a campaign to promote workplace policy and education on sun protection for outdoor workers. Primary outcome is adoption of formal policies and secondary outcomes are implementation of policy and sun protection practices by outdoor workers.

DETAILED DESCRIPTION:
Workers in the United States spend large amounts of time on the job, making the workplace a key venue for preventive health programs. A workplace risk that has received limited attention is sun protection, despite the fact 8% of the U.S. workforce (over 9 million workers) work outdoors. The investigators have demonstrated that sun safety education can promote sun protection at work. In this revised application, the investigators propose to systematically study a more comprehensive approach to workplace sun safety that goes beyond employee education to promote institutional change. The investigators will implement and evaluate a proactive campaign to change workplace sun protection policies and promote sun safety to managers rather than individual employees. The investigators will assess whether policy adoption alters organizational operations in public employers rather than the private employers examined in our previous research. The specific aims are to: a) create a campaign comprised of personal contacts, printed materials, and Internet tools and resources (i.e., pubic health communication) to promote workplace sun protection policies to managers at public employers, b) evaluate the effectiveness of the campaign at promoting adoption and implementation of workplace sun protection policies, and c) assess whether policy adoption is associated in increases in workers' sun protection practices. An advisory board of public administrators and health experts has been constituted to advise the investigators on campaign and evaluation procedures. Analysis of public employers' existing policies and practices, additional in-depth interviews with public administrators, information design analysis, and usability testing will be conducted to develop an effective campaign. The campaign will be evaluated in a group-randomized, pretest-posttest controlled design. City and county governments in Colorado will serve as the unit of randomization and analysis. Interviews will be conducted with a sample of administrators at these public employers at baseline, interim posttest (n=6 per employer) and final posttest (n=5 per employer). In a subsequent four-year follow-up, surveys with employees and front line supervisors will assess employees' sun protection practices and workplace actions to support employee sun safety; (2) on-site observations of sun protection actions by the employers (e.g., posters, sunscreen, shade structures) will be documented; and (3) costs of implementing the policy campaign and induced employer costs will be tracked. Public employers will be studied because they employ a sizable number of outdoor workers (but results should generalize to for-profit companies). Outcomes will be evaluated at the employer, administrator, and employee levels. At the employer level, adoption of workplace sun protection policies at pretest and each posttest will be assessed with a protocol for coding written workplace policies (primary outcome measure) that demonstrated high reliability in a pilot study. At the administrator level, policy implementation (secondary outcome), theoretical mediators of adoption and implementation, and individual, organizational, political decision making and program variables that might moderate change will be measured in baseline, interim posttest (halfway through the intervention) and final posttest (end of intervention) surveys. At the employee level, analyses will compare the sun protection practices of employees between workplaces that received the intervention and controls and among workplaces that provided education and adopted policy, provided education only, and control workplaces. Analyses will also determine if the extent of sun protection actions by employers influences employees' sun safety practices. At the cost level, the economic evaluation will estimate the return on investment (i.e., comparison of the estimated program benefits to combined cost elements). The proposed study is significant and innovative because it provides critical information applicable to a wide range of industrial sectors with outdoor workers on a workplace risk that has received scant attention. Determining the effectiveness and return on investment of prevention programs is essential for national and local resource investment.

ELIGIBILITY:
Inclusion Criteria:

* A local government organization with employees who worked outdoors in at least one of the following service areas: public works, public safety, and parks and recreation,
* Having a full time executive,
* Having a population of at least 3000 residents,
* Being employed at a participating local government organization as a manager
* Being employed at a participating local government organization in a job requiring outdoor work at least part of the time.

Exclusion Criteria:

* Organization had participated in the authors' previous occupational sun protection project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Presence of a Sun Protection Policy for Outdoor Workers | From baseline and 2-year follow-up
  Project staff coded written workplace policy documents on the presence of 15 "content categories" in three domains: 1) environmental controls; 2) administrative procedures; and 3) personal protection practices. Presence of policy was defined as having one or more policy components present in the written workplace policy documents (value=1) versus no content components present (value=0).

SECONDARY OUTCOMES:
Workplace Actions on Occupational Sun Safety | 2-year follow-up
  Managers reported whether local government organization provided any of the following to employees (0=No, 1=Yes): sunscreen, wide-brimmed hats, sunglasses, long-sleeved work or uniform shirts, long work or uniform pants, temporary or permanent shade, adjusted works schedules to reduce time outdoor at midday, communication about sun protection with employees. Total number of actions performed at the local government organization was summed.
Change in Awareness of a Sun Protection Policy for Outdoor Workers | From baseline to 2-year follow-up
  Managers reported whether the local government organization had formal written policy, administrative procedure, or training standard on sun protection for its employees (0=No or Don't Know, 1=Yes).
Sun Protection Practices by Outdoor Workers | 4-year follow-up
  Employees who work outdoors reported their frequency of taking the following actions to protect their skin from the sun (1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always): apply sunscreen with sun protection factor (SPF) of 15 or more, wear clothing specifically to protect skin from the sun such as long-sleeved shirts and pants, wear a hat with a brim, wear a hat with a wide-brim, wear sunglasses, limit exposure to the sun during the midday hours, and stay mostly in the shade. The frequency rating are averaged to form a composite sun protection score.
Change in Extent of Sun Protection Policy for Outdoor Workers | From baseline to 2-year follow-up
  Project staff coded written workplace policy documents on the presence of 15 "content categories" in three domains: 1) environmental controls; 2) administrative procedures; and 3) personal protection practices. Extent of policy was defined as the number of policy content components present in the written workplace policy documents (values=0 to 15).
Change in Strength of Sun Protection Policy for Outdoor Workers | From baseline to 2-year follow-up
  Project staff coded written workplace policy documents on the presence of 15 "content categories" in three domains: 1) environmental controls; 2) administrative procedures; and 3) personal protection practices. Extent of policy was defined as the sum of the strength scores (0=no advice; 1=recommended; 2=required) for each policy content component present in the written workplace policy documents (values=0 to 30).

CONTACTS AND LOCATIONS:
Overall Officials: David B Buller, PhD, Principal Investigator — Klein Buendel, Inc.
Locations (3):
- United States (3):
  - Kaiser Foundation Research Institute, Oakland, California
  - University of Colorado Denver, Aurora, Colorado
  - Klein Buendel, Inc., Golden, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walkosz BJ, Buller DB, Andersen PA, Wallis A, Buller MK, Scott MD. Factors Associated With Occupational Sun-Protection Policies in Local Government Organizations in Colorado. JAMA Dermatol. 2015 Sep;151(9):991-7. doi: 10.1001/jamadermatol.2015.0575. PMID 25993051
- [Background] Wallis A, Andersen PA, Buller DB, Walkosz B, Lui L, Buller M, Scott MD, Jenkins R. Adoption of sun safe workplace practices by local governments. J Public Health Manag Pract. 2014 Nov-Dec;20(6):608-16. doi: 10.1097/PHH.0000000000000026. PMID 24231670